CLINICAL TRIAL: NCT03278548
Title: Prospective, Randomized, Controlled, Double-blind, Multi-centre, Multinational Study on the Safety and Efficacy of 6% Hydroxyethyl Starch (HES) Solution Versus an Electrolyte Solution in Patients Undergoing Elective Abdominal Surgery
Brief Title: Safety and Efficacy of 6% Hydroxyethyl Starch (HES) Solution Versus an Electrolyte Solution in Patients Undergoing Elective Abdominal Surgery
Acronym: PHOENICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: B. Braun Melsungen AG (Industry); European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-1504; HE06-024-CP4 (Other: Fresenius Kabi)
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hypovolaemia Due to Acute Blood Loss
Keywords: HES; HES 130; Hydroxyethyl starch
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volulyte 6% (Experimental): Volulyte 6% solution for infusion
  Interventions: Drug: Volulyte 6%
- Ionolyte (Active Comparator): Ionolyte solution for infusion
  Interventions: Drug: Ionolyte

INTERVENTIONS:
Drug: Volulyte 6% — Solution for infusion
  Other Names: Hydroxyethyl starch 130/0.4
  Arms: Volulyte 6%
Drug: Ionolyte — Solution for infusion
  Other Names: Electrolyte solution
  Arms: Ionolyte

SUMMARY:
The aim of the study is to investigate the safety of a 6% HES (Hydroxyethyl Starch) solution (Volulyte 6%) versus an electrolyte solution (Ionolyte) in patients undergoing elective abdominal surgery.

ELIGIBILITY:
Inclusion:

* Male or female adult patients > 40 and ≤ 85 years of age. Women of child bearing potential must test negative on standard pregnancy test (urine or serum)
* Patients undergoing elective abdominal surgery with an expected blood loss of ≥ 500 ml
* ASA Physical Status II - III
* Signed written informed consent form

Exclusion:

* Hypersensitivity to the active substances or to any of the other excipients of the investigational medicinal products
* Body weight ≥ 140 kg
* Sepsis
* Burns
* Renal impairment (AKIN stage ≥ 1 or chronic) or acute and/or chronic renal replacement therapy
* Intracranial or cerebral haemorrhage
* Critically ill patients (typically admitted to the intensive care unit)
* Hyperhydration
* Pulmonary oedema
* Dehydration
* Hyperkalaemia
* Severe hypernatraemia
* Severe hyperchloraemia
* Severely impaired hepatic function
* Congestive heart failure
* Severe coagulopathy
* Organ transplant patients
* Metabolic alkalosis
* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)

Ages: 41 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2289 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Difference in mean estimated glomerular filtration rate (eGFR) (calculated from highest cystatin-C levels measured during post-operative days 1-3 (POD 1-3)) between the two treatment groups | post-operative days 1-3

SECONDARY OUTCOMES:
Renal function | until 1 year after surgery
Calculated red blood cell (RBC) loss | on post-operative day 3
Estimated intra-operative blood loss | end of surgery
Coagulation | until post-operative day 1
Inflammation | until post-operative day 1
Adverse events | until post-operative day 90
Major post-operative complications | until post-operative day 90
Mortality | 1 year
Composite of mortality and major post-operative complications (including renal) | until post-operative day 90
Total volume of administered investigational product | until 24 hours after investigational product treatment start
Fluid balance [Sum of volume of all intravenous medication (including investigational product and blood products) minus sum of volume of urine output (if available), drainage and estimated intra-operative blood loss] | until post-operative day 3
Heart Rate | until post-operative day 3
Body temperature | until post-operative day 3
Mean arterial pressure | until post-operative day 3, if available
Systolic arterial blood pressure | until end of surgery
Diastolic arterial blood pressure | until end of surgery
Central venous pressure (if available) | until end of surgery
Haemodynamics readings as required to determine volume responsiveness [at least one parameter (stroke volume, stroke volume variation, stroke volume index, pulse pressure variation, mean arterial pressure) has to be used to guide volume administration] | until 24 hours after investigational product treatment start
Partial pressure of carbon dioxide | until end of surgery
Partial pressure of oxygen | until end of surgery
Bicarbonate | until end of surgery
Arterial oxygen saturation | until end of surgery
Haemoglobin | until post-operative day 3
Haematocrit | until post-operative day 3
pH | until end of surgery
Base Excess | until end of surgery
Lactate | until post-operative day 3
Central venous oxygen saturation (if available) | until post-operative day 1
Serum sodium | until post-operative day 1
Serum potassium | until post-operative day 1
Serum calcium | until post-operative day 1
Serum chloride | until post-operative day 1
Length of stay in the hospital/intensive care unit | until post-operative day 90
Hours on mechanical ventilation | until post-operative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang F. Buhre, Prof. Dr. med., Study Chair — Department of Anesthesiology and Pain Management, Maastricht University, The Netherlands
Locations (61):
- Austria (2):
  - General Hospital of Barmherzige Brüder, Sankt Veit
  - Social Medical Center East - Donauspital, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Maria Middelares, Ghent
  - Jessa Ziekenhuis, Hasselt
- Croatia (3):
  - Clinical Hospital Sveti Duh, Zagreb
  - University Hospital Sisters of Mercy, Zagreb
  - University Hospital Zagreb, Zagreb
- Czechia (4):
  - Kolín Hospital, Kolín
  - Central Military Hospital Prague, Prague
  - General University Hospital in Prague, Prague
  - University Hospital Motol, Prague
- France (11):
  - CHU Angers, Angers
  - Hospital Centre Pierre Oudot, Bourgoin
  - CHRU Lille, Lille
  - Hospital Centre Montauban, Montauban
  - Montpellier University Hospital, Montpellier
  - AP-HP Paris (Salpêtrière), Paris
  - Hospital Saint-Antoine, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - University Hospital of Strasbourg, Strasbourg
  - Hospital Foch Suresnes, Suresnes
  - Hospital Jean Bernard, Valenciennes
- Germany (10):
  - Kliniken der Stadt Köln, Cologne
  - Carl-Thiem-Klinikum, Cottbus
  - Helios Amper-Klinikum, Dachau
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
  - University Hospital Marburg, Marburg
  - University Hospital Munich, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg AÖR, Oldenburg
  - Regio Klinikum Pinneberg GmbH, Pinneberg
- Netherlands (4):
  - Amsterdam Medical Centre, Amsterdam
  - Martini General Hospital Groningen, Groningen
  - University Medical Center Groningen, Groningen
  - University Medical Center (UMC) Maastricht, Maastricht
- Poland (9):
  - University Clinical Center Gdansk, Gdansk
  - Szpital Specjalistyczny im. Św. Łukasza, Gmina Końskie
  - Medical University of Silesia, Katowice
  - Wojewodzki Szpital Zespolony, Konin
  - Jagiollonian University Hospital Medical College, Krakow
  - Medical University of Lublin, Lublin
  - Karol Marcinkowski Medical University in Poznań, Poznan
  - University Hospital in Wroclaw, Wroclaw
  - Klinika Wiśniowa, Zielona Góra
- Romania (4):
  - Fundeni Clinical Institute 1, Bucharest
  - Fundeni Clinical Institute 2, Bucharest
  - University Hospital Elias Bucharest, Bucharest
  - Emergency county hospital Cluj, Cluj-Napoca
- Spain (11):
  - Barcelona Clinic Hospital, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - University Hospital General Del Elche, Elche
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Gregorio Marañon, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Quironsalud, Málaga
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia
  - Hospital Universitario Rio Hortega, Valladolid

REFERENCES:
- [Derived] Buhre W, Diaz-Cambronero O, Schaefer S, Novacek M, Domingo MS, Stessel B, Rodriguez-Perez A, Richter T, Rohe G, Cholley B, Gruenewald M, Kuiper G, Jaber S, de Korte D, Belda J, de Abreu MG, Baronica R, Scheeren T, Ferrando-Ortola C, Szczeklik W, Tomescu D, Vyzamal T, Gavranovic Z, Argente-Navarro MP, Mazzinari G, Thaler S, Garcia-Gregorio N, Vandenbrande J, Zlotnik D, Wittenstein J, Schmier S, Rohn S, Glasmacher C, Holler M, Jungheinrich C, Niess U, Sessler DI, Westphal M. Safety and efficacy of 6% hydroxyethyl starch in patients undergoing major surgery: The randomised controlled PHOENICS trial. Eur J Anaesthesiol. 2026 Jan 1;43(1):1-10. doi: 10.1097/EJA.0000000000002307. Epub 2025 Oct 24. PMID 41133731
- [Derived] Buhre W, de Korte-de Boer D, de Abreu MG, Scheeren T, Gruenewald M, Hoeft A, Spahn DR, Zarbock A, Daamen S, Westphal M, Brauer U, Dehnhardt T, Schmier S, Baron JF, De Hert S, Gavranovic Z, Cholley B, Vymazal T, Szczeklik W, Bornemann-Cimenti H, Soro Domingo MB, Grintescu I, Jankovic R, Belda J. Prospective, randomized, controlled, double-blind, multi-center, multinational study on the safety and efficacy of 6% Hydroxyethyl starch (HES) sOlution versus an Electrolyte solutioN In patients undergoing eleCtive abdominal Surgery: study protocol for the PHOENICS study. Trials. 2022 Feb 22;23(1):168. doi: 10.1186/s13063-022-06058-6. PMID 35193648
- [Derived] Chappell D, Jacob M. Should hydroxyethyl starch be banned? Lancet. 2018 Jul 14;392(10142):118. doi: 10.1016/S0140-6736(18)31174-7. No abstract available. PMID 30017128